CLINICAL TRIAL: NCT06534229
Title: Impact of Preoperative Endoscopic Ultrasound-guided Fine-needle Aspiration in Cholangiocarcinoma Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Other Study IDs: ROSC01
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Cholangiocarcinoma Patients
MeSH Terms: interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Endoscopic ultrasound-guided fine-needle aspiration — Endoscopic ultrasound-guided fine-needle aspiration for biopsy

SUMMARY:
Primary objective of this study is to evaluate the number of patients with positive LN detected by EUS and precluded from further surgical interventions.

Secondary objective of this study is to evaluate the EUS-related adverse events.

DETAILED DESCRIPTION:
Cholangiocarcinoma (CCA) is a rare malignancy originating from the bile duct epithelium. The incidence of CCA ranges from 0.5-2.5 cases per 100.000 people in West-European countries and 1.6 cases per 100.000 people in the United States of America. CCA is classified based on anatomical site and is divided into intrahepatic (iCCA), perihilar (pCCA) and distal (dCCA). Survival is limited, as CCA is often recognized in a relatively late stadium in which potential curative treatment is not an option anymore.

Currently, surgical resection is the only potentially curative treatment. The resectability of CCA depends on multiple factors: e.g. biliary extension, vascular involvement and presence of metastatic disease. Patients with metastatic disease, including both distant lymph nodes and metastases, are ineligible for surgical resection and palliative treatment should be initiated instead. Therefore, correct lymph node (N) staging is crucial. N staging depends on CCA subtype and differs between the 7th and 8th edition of The American Joint Committee on Cancer (AJCC) staging system. The most important difference between the two staging systems is the location of the regional (N1) versus distant lymph nodes (N2) in the 7th edition for pCCA and dCCA, while in the 8th edition distant N locations are considered M1 metastases and the number of lymph nodes determines the N stage. In both editions N locations in iCCA are subdivided for the left and right sided liver segments.The AJCC staging system is used to determine treatment and is correlated to survival. The 5-year survival for patients with regional or non-regional positive lymph nodes is worse compared to patients with negative lymph nodes.

To identify distant and lymph node metastases Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) is performed. However, it is difficult to accurately identify suspicious lymph nodes on both CT and MRI since sensitivity and specificity is 61% and 88% respectively for CT and 64% and 68% respectively for MRI. To assess lymph node staging more accurately, Endoscopic Ultrasound (EUS) with Fine Needle Aspiration (FNA) might be of added value. Only a few retrospective studies have described the yield of preoperative EUS for CCA. It is clear that EUS is an effective technique for lymph node staging for CCA, but data is inconsistent about the exact value and impact of EUS on clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a patient must meet the following criteria:

* Suspected resectable CCA
* Patient underwent EUS preoperatively

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from inclusion:

• History of treated CCA

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients are included retrospectively. Likely, a total of 100 patients are included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-25 (Estimated); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
Lymph node detection by EUS | 2024 - 2026
  Primary objective of this study is to evaluate the number of patients with positive LN detected by EUS and precluded from further surgical interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- AIG Hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No